CLINICAL TRIAL: NCT01251614
Title: A Multicenter, Randomized, Double-dummy, Double-blind Study Evaluating Two Doses of Adalimumab Versus Methotrexate (MTX) in Pediatric Subjects With Chronic Plaque Psoriasis (Ps)
Brief Title: A Double Blind Study in Pediatric Subjects With Chronic Plaque Psoriasis, Studying Adalimumab vs. Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M04-717; 2009-013072-52 (EudraCT Number)
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-08

CONDITIONS: Plaque Psoriasis
Keywords: Randomized; Double-blind; Chronic plaque psoriasis; Pediatric
MeSH Terms: interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Adalimumab 0.4 mg/kg (Experimental): In Period A participants received a single subcutaneous loading dose of adalimumab 0.4 mg/kg (up to a maximum of 20 mg) at Week 0 followed by every other week dosing beginning at Week 1. To maintain the blind, participants also received weekly dosing of methotrexate placebo tablets. Participants who were non-responders in Period A entered Period D directly and received open-label adalimumab at 0.8 mg/kg eow for up to 52 weeks. Participants who responded in Period A entered the Treatment Withdrawal Phase (Period B) for up to 36 weeks. Participants who experienced a loss of disease control in Period B entered the Re-treatment Phase (Period C) and received blinded adalimumab 0.4 mg/kg eow for 16 weeks. Participants who completed Period B with no loss of disease control entered Period D and were observed off study medication for up to 52 weeks. Participants who completed Period C entered Period D for an additional 52 weeks of treatment with blinded adalimumab 0.4 mg/kg eow.
  Interventions: Biological: Adalimumab; Drug: Placebo to Methotrexate
- Adalimumab 0.8 mg/kg (Experimental): In Period A participants received a single subcutaneous loading dose of adalimumab 0.8 mg/kg (up to a maximum of 40 mg) at Week 0 followed by every other week dosing beginning at Week 1. To maintain the blind, participants also received weekly dosing of methotrexate placebo tablets. Participants who were non-responders in Period A entered Period D directly and received open-label adalimumab at 0.8 mg/kg eow for up to 52 weeks. Participants who responded in Period A entered the Treatment Withdrawal Phase (Period B) for up to 36 weeks. Participants who experienced a loss of disease control in Period B entered the Re-treatment Phase (Period C) and received blinded adalimumab 0.8 mg/kg eow for 16 weeks. Participants who completed Period B with no loss of disease control entered Period D and were observed off study medication for up to 52 weeks. Participants who completed Period C entered Period D for an additional 52 weeks of treatment with blinded adalimumab 0.8 mg/kg eow.
  Interventions: Biological: Adalimumab; Drug: Placebo to Methotrexate
- Methotrexate (Active Comparator): Participants received 0.1 mg/kg methotrexate at Baseline (Week 0), and up to 0.4 mg/kg weekly (maximum dose of 25 mg/week) in Period A. Participants also received adalimumab placebo as a single subcutaneous loading dose at Week 0, followed by every other week (eow) dosing from Week 1. Participants who were non-responders in period A entered Period D directly and received open-label adalimumab at 0.8 mg/kg eow for up to 52 weeks. Participants who responded in Period A entered the Treatment Withdrawal Phase (Period B) for up to 36 weeks. Participants who experienced a loss of disease control in Period B entered the Re-treatment Phase (Period C) and received blinded adalimumab 0.8 mg/kg eow for 16 weeks. Participants who completed Period B with no loss of disease control entered Period D and were observed off study medication for up to 52 weeks. Participants who completed Period C entered Period D for an additional 52 weeks of treatment with blinded adalimumab 0.8 mg/kg eow.
  Interventions: Drug: Methotrexate; Biological: Placebo to Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab by subcutaneous injection every other week (eow)
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 0.4 mg/kg; Adalimumab 0.8 mg/kg
Drug: Methotrexate — Methotrexate 0.1 mg/kg at Week 0 and up to 0.4 mg/kg per week (maximum dose of 25 mg/week) orally.
  Arms: Methotrexate
Biological: Placebo to Adalimumab — A single subcutaneous loading dose at Week 0 followed by eow dosing beginning at Week 1.
  Arms: Methotrexate
Drug: Placebo to Methotrexate — Orally once a week
  Arms: Adalimumab 0.4 mg/kg; Adalimumab 0.8 mg/kg

SUMMARY:
This study will compare how well adalimumab works versus methotrexate (MTX) in children with moderate to severe psoriasis in the short term. It will also study how safe and how well adalimumab works in the long term and how long disease response can be maintained after stopping therapy.

DETAILED DESCRIPTION:
The study had a 30-day screening period and a multi-period study design, as described below:

Period A - Primary Treatment Phase: Participants were randomized to receive adalimumab 0.8 mg/kg, adalimumab 0.4 mg/kg, or MTX in 1:1:1 ratio for 16 weeks.

Period B - Treatment Withdrawal Phase: Responders were withdrawn from active treatment and monitored for loss of disease control for up to 36 weeks.

Period C - Re-Treatment Phase: Participants who had experienced loss of disease control in Period B were re-treated with adalimumab for 16 weeks.

Period D - Long-Term Follow-Up Phase: Participants received adalimumab or were observed off-treatment (if disease remained under control) for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 4 years and < 18 years of age;
2. Subject weighs ≥ 13 kg;
3. Subject must have failed to respond to topical therapy;
4. Subject must need systemic treatment to control his/her disease and meet one of the following:

   * Physician's Global Assessment (PGA) ≥ 4
   * Body surface area (BSA) involved > 20%
   * Very thick lesions with BSA > 10%
   * Psoriasis Area and Severity Index (PASI) > 20
   * PASI > 10 and at least one of the following:

     * Active psoriatic arthritis unresponsive to non-steroid anti-inflammatory drugs (NSAIDs)
     * Clinically relevant facial involvement
     * Clinically relevant genital involvement
     * Clinically relevant hand and/or foot involvement
     * Children's Dermatology Life Quality Index (CDLQI) > 10
5. If subject is < 12 years of age and resides in a geographic region where heliotherapy is practical, subject must have failed to respond, be intolerant, or have a contraindication to heliotherapy, or is not a suitable candidate for heliotherapy;
6. If ≥ 12 years of age, subject must have failed to respond, be intolerant, or have a contraindication to phototherapy, or is not a suitable candidate for phototherapy;
7. Subject must have a clinical diagnosis of psoriasis for at least 6 months as determined by the subject's medical history and confirmation of diagnosis through physical examination by the Investigator;
8. Subject must have stable plaque psoriasis for at least 2 months prior to Baseline

Exclusion Criteria:

1. Prior biologic use other than prior treatment with etanercept;
2. Treatment with etanercept therapy within 4 weeks prior to the Baseline visit; 3. Methotrexate (MTX) use within the past year or prior MTX use at any time where the subject did not respond, or did not tolerate MTX;

4. Contraindication for treatment with MTX during the study; 5. Erythrodermic psoriasis, generalized or localized pustular psoriasis, medication-induced or medication exacerbated psoriasis or new onset guttate psoriasis; 6. Infection(s) requiring treatment with intravenous (IV) anti-infectives within 30 days prior to the Baseline Visit or oral anti-infectives within 14 days prior to the Baseline Visit; 7. Treatment of psoriasis with topical therapies such as corticosteroids, vitamin D analogs, or retinoids within 7 days prior to the Baseline visit; 8. Treatment of psoriasis with ultraviolet (UV)B phototherapy, excessive sun exposure, or the use of tanning beds within 7 days prior to the Baseline visit; 9. Treatment of psoriasis with ultraviolet A with psoralen (PUVA) phototherapy, non-biologic systemic therapies for the treatment of psoriasis, or systemic therapies known to improve psoriasis within 14 days prior to the Baseline visit.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Williams, MD, Study Director — AbbVie

REFERENCES:
- [Result] Papp K, Thaci D, Marcoux D, Weibel L, Philipp S, Ghislain PD, Landells I, Hoeger P, Kotkin C, Unnebrink K, Seyger M, Williams D. Efficacy and safety of adalimumab every other week versus methotrexate once weekly in children and adolescents with severe chronic plaque psoriasis: a randomised, double-blind, phase 3 trial. Lancet. 2017 Jul 1;390(10089):40-49. doi: 10.1016/S0140-6736(17)31189-3. Epub 2017 May 4. PMID 28478975
- [Derived] Horneff G, Seyger MMB, Arikan D, Kalabic J, Anderson JK, Lazar A, Williams DA, Wang C, Tarzynski-Potempa R, Hyams JS. Safety of Adalimumab in Pediatric Patients with Polyarticular Juvenile Idiopathic Arthritis, Enthesitis-Related Arthritis, Psoriasis, and Crohn's Disease. J Pediatr. 2018 Oct;201:166-175.e3. doi: 10.1016/j.jpeds.2018.05.042. Epub 2018 Jul 25. PMID 30054164
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 38 sites in Belgium, Canada, Chile, Czech Republic, Germany, Hungary, Italy, Mexico, Netherlands, Poland, Spain, Switzerland, and Turkey.
Pre-assignment Details: Participants were randomized to receive adalimumab 0.8 mg/kg, adalimumab 0.4 mg/kg, or methotrexate (MTX) in a 1:1:1 ratio and were stratified according to prior history of etanercept treatment.
Period: Overall Study
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Started | 37 | 39 | 38
Entered Period B | 13 (Only participants who were responders at Week 16 (Period A) entered the Treatment Withdrawal Phase) | 18 (Only participants who were responders at Week 16 (Period A) entered the Treatment Withdrawal Phase) | 23 (Only participants who were responders at Week 16 (Period A) entered the Treatment Withdrawal Phase)
Entered Period C | 8 (Only participants who experienced loss of disease control in Period B entered the Re-Treatment Phase) | 11 (Only participants who experienced loss of disease control in Period B entered the Re-Treatment Phase) | 19 (Only participants who experienced loss of disease control in Period B entered the Re-Treatment Phase)
Entered Period D | 36 (Long-Term Follow-Up Phase (52 Weeks)) | 36 (Long-Term Follow-Up Phase (52 Weeks)) | 36 (Long-Term Follow-Up Phase (52 Weeks))
Completed | 34 | 26 | 30
Not Completed | 3 | 13 | 8
Not completed — Adverse Event | 1 | 0 | 1
Not completed — Lack of Efficacy | 1 | 9 | 4
Not completed — Clearing of Psoriatic Lesions | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Loss of Disease Control | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg | Total
Number analyzed (Participants) | 37 | 39 | 38 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (3.49) | 12.6 (4.43) | 13.0 (3.29) | 13.0 (3.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 21 | 65
  Male | 11 | 21 | 17 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34 | 34 | 35 | 103
  Black | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 5
  American Indian/Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0
  Other | 1 | 2 | 2 | 5
  Mutli Race | 0 | 1 | 0 | 1
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: units on a scale] — PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  units on a scale | 19.2 (10.02) | 16.9 (5.76) | 18.9 (10.03) | 18.3 (8.78)
Physician's Global Assessment of Psoriasis [Count of Participants; unit: Participants] — The PGA is a 6-point scale used to measure the severity of disease using the following categories: 0 (Cleared): No scaling, erythema, or plaque elevation; 1 (Minimal): Occasional fine scale over < 5% of lesions, faint erythema, minimal plaque elevation; 2 (Mild): Fine scale, light red coloration, mild plaque elevation; 3 (Moderate): Course scale, moderate red coloration, moderate plaque elevation; 4 (Marked): Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation; 5 (Severe): Very thick tenacious scale, dusky to deep red coloration, severe plaque elevation.
  Participants
    Cleared | 0 | 0 | 0 | 0
    Minimal | 0 | 1 | 0 | 1
    Mild | 1 | 3 | 3 | 7
    Moderate | 19 | 18 | 17 | 54
    Marked | 17 | 15 | 17 | 49
    Severe | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI) 75 Response at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 75 response is defined as at least a 75% reduction (improvement) from Baseline in PASI score at Week 16.
Time Frame: Baseline and Week 16
Population: Non-responder imputation was used, the analysis was conducted in the intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Groups:
- Methotrexate: Participants received 0.1 mg/kg methotrexate at Baseline (Week 0), and up to 0.4 mg/kg weekly (maximum dose of 25 mg/week) in Period A. Participants also received adalimumab placebo as a single subcutaneous loading dose at Week 0, followed by every other week (eow) dosing from Week 1.
- Adalimumab 0.4 mg/kg: In Period A participants received a single subcutaneous loading dose of adalimumab 0.4 mg/kg (up to a maximum of 20 mg) at Week 0 followed by every other week dosing beginning at Week 1. To maintain the blind, participants also received weekly dosing of methotrexate placebo tablets.
- Adalimumab 0.8 mg/kg: In Period A participants received a single subcutaneous loading dose of adalimumab 0.8 mg/kg (up to a maximum of 40 mg) at Week 0 followed by every other week dosing beginning at Week 1. To maintain the blind, participants also received weekly dosing of methotrexate placebo tablets.
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants | 32.4 | 43.6 | 57.9
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; The a priori defined order of the statistical hypotheses was as follows: 1. Superiority of adalimumab 0.8 mg/kg versus MTX for the percentage of participants achieving a ≥ PASI 75 response at Week 16. 2. Superiority of adalimumab 0.8 mg/kg versus MTX, for the percentage of participants achieving a PGA cleared or minimal at Week 16. This order was adhered to for confirmatory testing, all statistical tests were at a level of significance of 5% and the overall type I error was preserved; Test type: Superiority or Other; p = 0.027, Chi-squared; Difference = -25.5, 95% CI 2-sided [-47.2 to -3.7]

2. Primary Outcome: Percentage of Participants Achieving a Physician's Global Assessment of Disease Activity (PGA) of "Cleared" (0) or "Minimal" (1) at Week 16
Description: The PGA is a 6-point scale used to measure the severity of disease at the time of the evaluation. The degree of overall lesion severity was evaluated using the following categories:
  * 0 (Cleared): No evidence of scaling, erythema, or plaque elevation;
  * 1 (Minimal): Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation;
  * 2 (Mild): Fine scale dominates, light red coloration, mild plaque elevation;
  * 3 (Moderate): Course scale dominates, moderate red coloration, moderate plaque elevation;
  * 4 (Marked): Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation;
  * 5 (Severe): Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation.
  The percentage of participants achieving a score of clear (0) or minimal (1) is reported.
Time Frame: Week 16
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants | 40.5 | 41.0 | 60.5
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.083, Chi-squared; Difference = -20.0, 95% CI 2-sided [-42.2 to 2.2]

3. Secondary Outcome: Percentage of Participants Who Achieved a PASI 90 Response at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  A PASI 90 response is at least a 90% reduction (improvement) from Baseline in PASI score at Week 16.
Time Frame: Baseline and Week 16
Population: Non-responder imputation was used, the analysis was conducted in the intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants | 21.6 | 30.8 | 28.9
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; Statistical comparisons for the ranked secondary endpoints were carried out in hierarchical order. All statistical tests were 2-sided with the significance level of 5%. Statistically significant results (p-value ≤ 0.05) must have been achieved for a comparison in the higher rank in order to initiate the next comparison in the lower rank; Test type: Superiority or Other; p = 0.466, Chi-squared; Difference = -7.3, 95% CI 2-sided [-26.9 to 12.3]

4. Secondary Outcome: Percentage of Participants Who Achieved a PASI 100 Response at Week 16
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  A PASI 100 response is a 100% reduction (improvement) from Baseline in PASI score at Week 16.
Time Frame: Baseline and Week 16
Population: Non-responder imputation was used, the analysis was conducted in the intent-to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants | 2.7 | 10.3 | 18.4
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.056, Fisher Exact; Difference = -15.7, 95% CI 2-sided [-29.1 to -2.3]

5. Secondary Outcome: Change From Baseline in the Children's Dermatology Life Quality Index (CDLQI) Score at Week 16
Description: The Children's Dermatology Life Quality Index (CDLQI) is a 10-item questionnaire to measure the quality of life in children aged from 4 to 16 years. Each question is scored from 0 (not at all) to 3 (very much). The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
Time Frame: Baseline and Week 16
Population: Last observation carried forward (LOCF) imputation was used, the analysis was conducted in the intent-to-treat (ITT) population; only participants with Baseline and at least one post-baseline value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 36 | 38 | 38
units on a scale | -5.0 (7.11) | -4.9 (6.16) | -6.6 (6.22)
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.304, ANOVA; Difference = 1.61, 95% CI 2-sided [-1.48 to 4.70]

6. Secondary Outcome: Change From Baseline in the Pediatric Quality of Life Inventory (PedsQL) Score at Week 16
Description: The PedsQL Measurement Model measures health-related quality of life (HRQOL) in children and adolescents. The 23-item PedsQL Generic Core Scale includes Physical, Emotional, Social, School Functioning dimensions. Each item is scored from 0 (never) to 4 (almost always). Items are reversed scored and linearly transformed to a 0-100 scale, so that higher scores indicate better HRQOL; the total score therefore ranges from 0 (worst) to 100 (best).
Time Frame: Baseline and Week 16
Population: LOCF imputation was used, the analysis was conducted in the intent-to-treat (ITT) population; only participants with Baseline and at least one post-baseline value are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 38 | 38
units on a scale | 1.9 (10.41) | 9.5 (12.25) | 10.8 (15.38)
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.005, ANOVA; Difference = -8.88, 95% CI 2-sided [-14.94 to -2.82]

7. Secondary Outcome: Percentage of Participants Achieving a PGA of "Cleared" (0) or "Minimal" (1) Upon Re-Treatment in Period C
Description: The PGA is a 6-point scale used to measure the severity of disease at the time of the evaluation. The degree of overall lesion severity was evaluated using the following categories: 0 (Cleared): No evidence of scaling, erythema, or plaque elevation; 1 (Minimal): Occasional fine scale over < 5% of lesions, faint erythema, minimal plaque elevation; 2 (Mild): Fine scale dominates, light red coloration, mild plaque elevation; 3 (Moderate): Course scale dominates, moderate red coloration, moderate plaque elevation; 4 (Marked): Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation; 5 (Severe): Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation. The percentage of participants achieving a score of clear (0) or minimal (1) is reported.
Time Frame: Period C, Week 16
Population: Non-responder imputation was used, the analysis was conducted in the ITT population who entered Period C.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 8 | 11 | 19
percentage of participants | 62.5 | 27.3 | 52.6
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.4 mg/kg vs Adalimumab 0.8 mg/kg; The difference between the combined adalimumab 0.8 mg/kg + MTX groups versus the adalimumab 0.4 mg/kg group. Statistical comparisons for the ranked secondary endpoints were carried out in hierarchical order. All statistical tests were to be 2-sided with the significance level of 5%. Statistically significant results (P value ≤ 0.05) must have been achieved for a comparison in the higher rank in order to initiate the next comparison in the lower rank; Test type: Superiority or Other; p = 0.113, Chi-squared; Difference = -28.3, 95% CI 2-sided [-60.6 to 4.0]

8. Secondary Outcome: Time to Loss of Disease Control for Participants Who Entered Period B
Description: Loss of disease control was defined as a worsening of PGA scores in comparison to Week 16 of Period A by at least 2 grades after treatment withdrawal. The PGA is a 6-point scale used to measure the severity of disease at the time of the evaluation. Scores range from 0 (no evidence of scaling, erythema, or plaque elevation) to 5 (very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation).
  Participants who did not lose disease control in period B continued off drug into period D and were observed off-drug until they finally lost disease control or until the end of the 52 weeks of period D.
Time Frame: Period B (36 weeks) and Period D (52 weeks)
Population: This analysis was conducted in the ITT population who entered period B, no imputation was used.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 13 | 18 | 23
days | 184 [84 to 335] | 217 [56 to 551] | 118 [79 to 194]
Statistical Analysis 1: Comparison: Methotrexate vs Adalimumab 0.8 mg/kg; Statistical comparisons for the ranked secondary endpoints were carried out in hierarchical order. All statistical tests were 2-sided with the significance level of 5%. Statistically significant results (P value ≤ 0.05) must have been achieved for a comparison in the higher rank in order to initiate the next comparison in the lower rank; Test type: Superiority or Other; p = 0.343, Log Rank; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.66 to 3.17]
Statistical Analysis 2: Comparison: Adalimumab 0.4 mg/kg vs Adalimumab 0.8 mg/kg; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.276, Log Rank; Hazard Ratio (HR) = 1.51, 95% CI 2-sided [0.71 to 3.21]

9. Secondary Outcome: Percentage of Participants Achieving a PGA of "Cleared" (0) or "Minimal" (1) Over Time
Description: The PGA is a 6-point scale used to measure the severity of disease at the time of the evaluation. The degree of overall lesion severity was evaluated using the following categories: 0 (Cleared): No evidence of scaling, erythema, or plaque elevation; 1 (Minimal): Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation; 2 (Mild): Fine scale dominates, light red coloration, mild plaque elevation; 3 (Moderate): Course scale dominates, moderate red coloration, moderate plaque elevation; 4 (Marked): Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation; 5 (Severe): Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation. The percentage of participants achieving a score of clear (0) or minimal (1) is reported.
Time Frame: Period A, Weeks 4, 8 and 11, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 8.1 | 20.5 | 28.9
  Period A, Week 8 | 8.1 | 35.9 | 44.7
  Period A, Week 11 | 18.9 | 30.8 | 47.4
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 0.0 | 0.0 | 0.0
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | 62.5 | 27.3 | 52.6
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 30.6 | 19.4 | 38.9
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | 77.8 | 38.9 | 50.0
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 69.4 | 50.0 | 63.9
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | 69.4 | 50.0 | 61.1
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 75.0 | 50.0 | 55.6

10. Secondary Outcome: Percentage of Participants Achieving a PGA of "Cleared" (0) Over Time
Description: The PGA is a 6-point scale used to measure the severity of disease at the time of the evaluation. The degree of overall lesion severity was evaluated using the following categories: 0 (Cleared): No evidence of scaling, erythema, or plaque elevation; 1 (Minimal): Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation; 2 (Mild): Fine scale dominates, light red coloration, mild plaque elevation; 3 (Moderate): Course scale dominates, moderate red coloration, moderate plaque elevation; 4 (Marked): Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation; 5 (Severe): Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation.
  The percentage of participants achieving a score of clear (0) is reported.
Time Frame: Period A, Weeks 4, 8, 11 and 16, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 0.0 | 2.6 | 2.6
  Period A, Week 8 | 0.0 | 12.8 | 5.3
  Period A, Week 11 | 0.0 | 10.3 | 10.5
  Period A, Week 16 | 8.1 | 12.8 | 18.4
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 0.0 | 0.0 | 0.0
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | 25.0 | 9.1 | 15.8
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 8.3 | 5.6 | 11.1
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | 25.0 | 11.1 | 25.0
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 33.3 | 16.7 | 22.2
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | 33.3 | 16.7 | 27.8
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 41.7 | 25.0 | 25.0

11. Secondary Outcome: Percentage of Participants Who Achieved a PASI 50 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  A PASI 50 response is at least a 50% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline, Period A, Weeks 4, 8, 11 and 16, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 16.2 | 41.0 | 52.6
  Period A, Week 8 | 40.5 | 56.4 | 65.8
  Period A, Week 11 | 51.4 | 61.5 | 71.1
  Period A, Week 16 | 54.1 | 66.7 | 78.9
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 62.5 | 90.9 | 52.6
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | 87.5 | 90.9 | 89.5
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 52.8 | 63.9 | 75.0
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | 91.7 | 69.4 | 88.9
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 88.9 | 72.2 | 86.1
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | 91.7 | 63.9 | 83.3
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 91.7 | 66.7 | 77.8

12. Secondary Outcome: Percentage of Participants Who Achieved a PASI 75 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  A PASI 75 response is at least a 75% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline, Period A, Weeks 4, 8, and 11, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 0.0 | 15.4 | 23.7
  Period A, Week 8 | 13.5 | 38.5 | 47.4
  Period A, Week 11 | 21.6 | 43.6 | 60.5
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 37.5 | 18.2 | 21.1
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | 75.0 | 54.5 | 78.9
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 30.6 | 27.8 | 50.0
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | 86.1 | 50.0 | 61.1
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 80.6 | 58.3 | 77.8
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | 77.8 | 52.8 | 75.0
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 86.1 | 47.2 | 72.2

13. Secondary Outcome: Percentage of Participants Who Achieved a PASI 90 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  A PASI 90 response is at least a 90% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline, Period A, Weeks 4, 8 and 11, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 0.0 | 5.1 | 5.3
  Period A, Week 8 | 2.7 | 20.5 | 23.7
  Period A, Week 11 | 2.7 | 28.2 | 28.9
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 0.0 | 0.0 | 10.5
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | 62.5 | 27.3 | 57.9
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 25.0 | 16.7 | 36.1
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | 63.9 | 36.1 | 38.9
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 55.6 | 33.3 | 41.7
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | 55.6 | 36.1 | 47.2
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 66.7 | 33.3 | 44.4

14. Secondary Outcome: Percentage of Participants Who Achieved a PASI 100 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
  A PASI 100 response is a 100% reduction (improvement) from Baseline in PASI score.
Time Frame: Baseline, Period A, Weeks 4, 8, and 11, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: Non-responder imputation was used, the analysis was conducted in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 0.0 | 0.0 | 2.6
  Period A, Week 8 | 0.0 | 5.1 | 5.3
  Period A, Week 11 | 0.0 | 5.1 | 10.5
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 0.0 | 0.0 | 0.0
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | 25.0 | 9.1 | 15.8
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 8.3 | 5.6 | 11.1
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | 13.9 | 11.1 | 25.0
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 27.8 | 13.9 | 19.4
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | 30.6 | 13.9 | 22.2
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 41.7 | 25.0 | 22.2

15. Secondary Outcome: Percent Change From Baseline in PASI Score Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
Time Frame: Baseline, Period A, Weeks 4, 8, 11 and 16, Period C, Weeks 0 and 16, Period D, Weeks 0, 16, 28, 40 and 52
Population: LOCF imputation was used, the analysis was conducted in the intent-to-treat (ITT) population.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percent change
  Period A, Week 4 | -14.0 (36.71) | -36.9 (38.62) | -48.3 (33.96)
  Period A, Week 8 | -30.6 (45.89) | -48.8 (44.74) | -60.3 (35.98)
  Period A, Week 11 | -36.6 (51.69) | -51.4 (50.19) | -62.8 (38.02)
  Period A, Week 16 | -42.8 (54.24) | -52.4 (51.79) | -65.6 (39.44)
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | -59.0 (20.61) | -65.3 (12.16) | -45.8 (39.64)
  Period C, Week 16: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 16 | -87.1 (16.47) | -74.5 (17.79) | -69.3 (69.79)
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | -41.8 (54.99) | -46.8 (49.27) | -61.5 (42.96)
  Period D, Week 16: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 16 | -82.3 (31.38) | -66.9 (33.51) | -74.5 (37.44)
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | -81.0 (35.86) | -65.8 (36.99) | -81.5 (22.06)
  Period D, Week 40: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 40 | -83.0 (31.94) | -64.6 (37.46) | -82.1 (23.99)
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | -86.3 (28.92) | -58.7 (53.21) | -80.1 (24.17)

16. Secondary Outcome: Change From Baseline in CDLQI Over Time
Description: as for outcome 5
Time Frame: Baseline, Period A, Weeks 4, and 8, Period C, Weeks 0 and 4, Period D, Weeks 0, 11, 28, and 52
Population: LOCF imputation was used, the analysis was conducted in the intent-to-treat (ITT) population with available data at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 36 | 38 | 38
units on a scale
  Period A, Week 4 | -2.9 (5.24) | -3.9 (5.22) | -4.9 (5.80)
  Period A, Week 8 | -4.0 (6.44) | -4.1 (6.29) | -5.5 (5.66)
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | -6.1 (4.55) | -4.7 (9.08) | -6.1 (6.92)
  Period C, Week 4: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 4 | -9.8 (3.92) | -5.5 (7.24) | -7.0 (6.63)
  Period D, Week 0: number analyzed (Participants) | 35 | 35 | 36
  Period D, Week 0 | -5.6 (7.55) | -5.5 (5.95) | -6.8 (6.70)
  Period D, Week 11: number analyzed (Participants) | 35 | 35 | 36
  Period D, Week 11 | -8.5 (5.37) | -6.8 (7.07) | -7.4 (6.21)
  Period D, Week 28: number analyzed (Participants) | 35 | 35 | 36
  Period D, Week 28 | -8.3 (5.93) | -6.8 (7.91) | -8.4 (6.72)
  Period D, Week 52: number analyzed (Participants) | 35 | 35 | 36
  Period D, Week 52 | -8.4 (6.08) | -6.6 (8.12) | -8.2 (6.75)

17. Secondary Outcome: Percentage of Participants With CDLQI = 0 Over Time
Description: The Children's Dermatology Life Quality Index (CDLQI) is a 10-item questionnaire to measure the quality of life in children aged from 4 to 16 years. Each question is scored from 0 (not at all) to 3 (very much). The CDLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired and a score of 0 indicates no impairment in quality of life.
Time Frame: Period A, Weeks 4, 8 and 16, Period C, Weeks 0 and 4, Period D, Weeks 0, 11, 28, and 52
Population: Non-responder imputation was used, the analysis was conducted in the intent to-treat (ITT) population.
Measure: Number; unit: percentage of participants
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
percentage of participants
  Period A, Week 4 | 5.4 | 5.1 | 10.5
  Period A, Week 8 | 10.8 | 12.8 | 5.3
  Period A, Week 16 | 10.8 | 20.5 | 23.7
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 0.0 | 36.4 | 21.1
  Period C, Week 4: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 4 | 12.5 | 36.4 | 31.6
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 16.7 | 22.2 | 27.8
  Period D, Week 11: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 11 | 25.0 | 16.7 | 33.3
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 30.6 | 22.2 | 30.6
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 41.7 | 16.7 | 33.3

18. Secondary Outcome: Time to PASI 50/75/90/100 Response in Period A
Description: Participants who did not have a response during Period A were censored.
Time Frame: Period A, 16 weeks
Population: Analysis was conducted in the intent to-treat (ITT) population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 39 | 38
days
  PASI 50 | 76 [56 to 112] | 55 [28 to 115] | 30 [28 to 77]
  PASI 75 | 116 [111 to NA] — Not estimable due to the low number of events | 107 [56 to NA] — Not estimable due to the low number of events | 59 [53 to NA] — Not estimable due to the low number of events
  PASI 90 | NA [112 to NA] — Not estimable due to the low number of events | NA [78 to NA] — Not estimable due to the low number of events | NA [76 to NA] — Not estimable due to the low number of events
  PASI 100 | NA [NA to NA] — Not estimable due to the low number of events | NA [NA to NA] — Not estimable due to the low number of events | NA [NA to NA] — Not estimable due to the low number of events

19. Secondary Outcome: Change From Baseline in PedsQL Over Time
Description: as for outcome 6
Time Frame: Baseline, Period A, Weeks 4 and 8, Period C, Weeks 0 and 4, Period D, Weeks 0, 11, 28, and 52
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 37 | 38 | 38
units on a scale
  Period A, Week 4: number analyzed (Participants) | 37 | 38 | 36
  Period A, Week 4 | -0.8 (11.75) | 4.9 (13.80) | 8.1 (11.95)
  Period A, Week 8 | 0.5 (10.18) | 7.0 (13.16) | 8.8 (15.45)
  Period C, Week 0: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 0 | 3.0 (10.45) | 8.9 (25.35) | 14.2 (20.25)
  Period C, Week 4: number analyzed (Participants) | 8 | 11 | 19
  Period C, Week 4 | 5.2 (11.08) | 11.6 (25.19) | 16.3 (17.35)
  Period D, Week 0: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 0 | 2.3 (10.93) | 9.4 (16.90) | 10.5 (15.86)
  Period D, Week 11: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 11 | 5.4 (10.36) | 12.8 (19.03) | 12.0 (16.13)
  Period D, Week 28: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 28 | 8.0 (13.40) | 14.5 (20.19) | 13.1 (16.23)
  Period D, Week 52: number analyzed (Participants) | 36 | 36 | 36
  Period D, Week 52 | 8.6 (13.93) | 14.0 (20.40) | 13.8 (15.36)

20. Secondary Outcome: Change From Baseline in the Children's Depression Inventory: Short (CDI:S)
Description: The CDI:S is a short 10-item self-rated symptom-oriented scale used to screen for depressive symptoms. CDI:S scores range from 0 to 100, with a lower score indicating fewer depressive symptoms.
Time Frame: Baseline, Period A, Weeks 4, 8, and 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg
Number analyzed (Participants) | 36 | 35 | 36
units on a scale
  Period A, Week 4: number analyzed (Participants) | 35 | 35 | 34
  Period A, Week 4 | 0.6 (8.85) | -1.0 (6.64) | -3.6 (5.86)
  Period A, Week 8: number analyzed (Participants) | 35 | 35 | 34
  Period A, Week 8 | 0.2 (5.26) | -1.5 (7.52) | -1.6 (5.52)
  Period A, Week 16: number analyzed (Participants) | 35 | 35 | 35
  Period A, Week 16 | -2.0 (5.88) | -3.3 (8.12) | -2.3 (6.29)

ADVERSE EVENTS:
Time Frame: Period A - up to 16 weeks; Period B - up to 36 weeks; Period C - up to 16 weeks; Period D - up to 52 weeks.
Groups:
- Period B: MTX/No Treatment: Participants initially randomized to methotrexate who responded in Period A were withdrawn from active therapy in Period B for up to 36 weeks.
- Period B: ADA 0.4 mg/kg/No Treatment: Participants initially randomized to adalimumab (ADA) 0.4 mg/kg who responded in Period A were withdrawn from active therapy in Period B for up to 36 weeks.
- Period B: ADA 0.8 mg/kg/No Treatment: Participants initially randomized to adalimumab (ADA) 0.8 mg/kg who responded in Period A were withdrawn from active therapy in Period B for up to 36 weeks.
- Period C: Adalimumab 0.4 mg/kg: Participants initially randomized to adalimumab 0.4 mg/kg with loss of disease control in Period B received adalimumab 0.4 mg/kg eow for up to 16 weeks in Period C.
- Period C: Adalimumab 0.8 mg/kg: Participants initially randomized to either methotrexate or adalimumab 0.8 mg/kg with loss of disease control in Period B received adalimumab 0.8 mg/kg eow for up to 16 weeks in Period C.
- Period D: Adalimumab 0.4 mg/kg: Participants received adalimumab 0.4 mg/kg eow for up to 52 weeks in Period D.
- Period D: Adalimumab 0.8 mg/kg: Participants received adalimumab 0.8 mg/kg eow for up to 52 weeks in Period D.
Arm/Group | Methotrexate | Adalimumab 0.4 mg/kg | Adalimumab 0.8 mg/kg | Period B: MTX/No Treatment | Period B: ADA 0.4 mg/kg/No Treatment | Period B: ADA 0.8 mg/kg/No Treatment | Period C: Adalimumab 0.4 mg/kg | Period C: Adalimumab 0.8 mg/kg | Period D: Adalimumab 0.4 mg/kg | Period D: Adalimumab 0.8 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/37 | 3/39 | 0/38 | 0/13 | 0/18 | 1/23 | 0/11 | 0/27 | 0/13 | 5/87
Other Adverse Events (participants affected / at risk) | 23/37 | 27/39 | 23/38 | 6/13 | 6/18 | 6/23 | 5/11 | 16/27 | 8/13 | 64/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=37) | Adalimumab 0.4 mg/kg (N=39) | Adalimumab 0.8 mg/kg (N=38) | Period B: MTX/No Treatment (N=13) | Period B: ADA 0.4 mg/kg/No Treatment (N=18) | Period B: ADA 0.8 mg/kg/No Treatment (N=23) | Period C: Adalimumab 0.4 mg/kg (N=11) | Period C: Adalimumab 0.8 mg/kg (N=27) | Period D: Adalimumab 0.4 mg/kg (N=13) | Period D: Adalimumab 0.8 mg/kg (N=87)
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye Naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=37) | Adalimumab 0.4 mg/kg (N=39) | Adalimumab 0.8 mg/kg (N=38) | Period B: MTX/No Treatment (N=13) | Period B: ADA 0.4 mg/kg/No Treatment (N=18) | Period B: ADA 0.8 mg/kg/No Treatment (N=23) | Period C: Adalimumab 0.4 mg/kg (N=11) | Period C: Adalimumab 0.8 mg/kg (N=27) | Period D: Adalimumab 0.4 mg/kg (N=13) | Period D: Adalimumab 0.8 mg/kg (N=87)
Abdominal Pain (Gastrointestinal disorders) | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 10
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 3
Asthenia (General disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 4
Injection Site Pain (General disorders) | 3 | 1 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Injection Site Reaction (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 5
Gastroenteritis (Infections and infestations) | 3 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 9
Lice Infestation (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 10 | 8 | 0 | 1 | 4 | 1 | 5 | 3 | 25
Oral Herpes (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Pharyngitis Streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 6 | 4 | 2 | 0 | 2 | 1 | 0 | 3 | 0 | 13
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Varicella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Joint Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 4
Headache (Nervous system disorders) | 4 | 7 | 6 | 1 | 2 | 1 | 0 | 3 | 1 | 22
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 0 | 2 | 0 | 2 | 1 | 1 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 4
Eczema Vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 4
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.